CLINICAL TRIAL: NCT04722822
Title: The HPV 9-10 Trial: Early Initiation of HPV Vaccination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-3006.cc; 1R01CA240649-01A1 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: HPV
MeSH Terms: interventions — Methods; Aging

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator and data analysis team will be blinded to the arms during analysis. Practices (unit of randomization) cannot be blinded; however patients who are subjects of the intervention are not aware of the group allocation of the practice in the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients attributed to practices recommending HPV at age 9-10 years of age (Experimental): Patients attributed to practices routinely recommending HPV vaccine starting at 9-10 years of age.
  Interventions: Behavioral: (Intervention) Recommending HPV vaccine for patients 9-10 years of age
- Patients attributed to practices recommending HPV at age 11-12 years of age (Active Comparator): Patients attributed to practices routinely recommending HPV vaccine starting at 11-12 years of age.
  Interventions: Behavioral: (Control) Recommending HPV vaccine for patients 11-12 years of age

INTERVENTIONS:
Behavioral: (Intervention) Recommending HPV vaccine for patients 9-10 years of age — Practices are randomized to receive training on how to recommend HPV vaccine, including both standardized communication strategies and strategies for switching from 11-12 years to 9-10 years including: challenges with 11-12 strategy, long-term immunity, success of other practices and tips to help standardize to age 9-10. Trainings will be a combination of online and in-person or virtual. Annual trainings will be offered and providers will receive Maintenance of Certification credits (MOC) for participating. Providers will routinely recommend HPV starting at age 9 for all patients -- which is already approved for this vaccine but is not routinely recommended at age 9 years.
  Arms: Patients attributed to practices recommending HPV at age 9-10 years of age
Behavioral: (Control) Recommending HPV vaccine for patients 11-12 years of age — Control practices will receive a training on standardized communication for HPV vaccine including: using strong recommendations, using presumptive recommendation, providing specific phrases to use with parents, answering common questions and, HPV vaccine as a cancer prevention. Annual trainings will be offered and providers will receive professional development credit (MOC).
  Arms: Patients attributed to practices recommending HPV at age 11-12 years of age

SUMMARY:
Every year, thousands of Americans die from cancers related to human papillomavirus (HPV). The vast majority of those deaths could be prevented with a safe and effective vaccine, yet many parents choose not have their children vaccinated when it is recommended at age 11 or 12. In this study, we will examine in a randomized trial whether earlier initiation of the vaccine at age 9-10 years will result in less parental refusal and higher rates of full vaccination at younger ages, before early sexual activity begins.

DETAILED DESCRIPTION:
The burden of Human Papillomavirus (HPV)-related disease in the US is substantial. A safe and effective vaccine has been available for >10 years, yet the current rate of completion for the HPV series is only 49% for U.S.13-17 year olds. The Advisory Committee on Immunization Practices (ACIP) recommends routine HPV vaccination at age 11-12 years (yrs), but states that the vaccine "can be given starting at age 9 years." Currently, the majority of pediatricians begin recommending the vaccine at ages 11-12 yrs, however, a recent retrospective study showed that on-time completion rates for HPV vaccine were much higher when the vaccine series was initiated at ages 9-10 compared to ages 11-12 (adjusted odds ratio, 12.8).

HPV vaccine should be given prior to sexual activity which occurs earlier than 13 yrs for many teens. There are compelling reasons to think that earlier initiation of vaccination at ages 9-10 might result in higher rates of acceptance of the vaccine and earlier series completion. First, many parents refuse HPV vaccine because they have concerns that vaccination could result in higher promiscuity in early adolescents if the vaccine is discussed in the context of sexuality. Initiation at 9-10 yrs, when few providers discuss sex, could put the focus squarely on cancer prevention, decreasing vaccine refusal. Second, three vaccines are recommended at the 11-12 yr visit, but many parents/adolescents are unwilling to receive all three at one visit. When one of the vaccines is delayed, it is almost always HPV vaccine. Initiation at 9-10 yrs when no other vaccines are given could result in less deferral of vaccination to mid-adolescence and higher rates of vaccination prior to early sexual activity. Finally, initiation at age 9-10 years has been shown to be feasible and, in an observational study, to result in higher rates of on-time series completion.

Therefore, we plan to test the effectiveness of shifting initiation of HPV vaccine to 9-10 yrs in a randomized pragmatic trial. Our Specific Aims are to: SA 1: Recruit practices in two states (Colorado and California), randomize in a balanced fashion to recommending HPV vaccine at ages 9-10 yrs or 11-12 yrs and provide standardized training to both arms. SA 2: Conduct a trial to assess effectiveness of early initiation on the primary outcome of age at HPV series completion; secondary outcomes will examine HPV series completion by age 13 and age at HPV series initiation. SA 3: Examine the effect of earlier initiation on length of time for HPV vaccine discussions and on parent/provider communication about HPV vaccine via audio-taping of visits, audio-elicitation interviews with parents and structured interviews with providers and clinic staff.

If earlier HPV initiation is successful in promoting higher HPV series completion by 13 yrs, this intervention could be rapidly disseminated and would have the potential to prevent thousands of cases of HPV-related cancers, their attendant morbidity and mortality as well as the costs of screening, diagnosis and treatment for these cancers yearly.

ELIGIBILITY:
Practices:

Inclusion Criteria:

* Practices in Metro Denver, Colorado and Metro Los Angeles, California (specifically UCLA medical clinics and clinics affiliated with Children's Hospital of Orange County)
* Practices that have at least 60% of providers agree to participate
* Practices do not currently recommend HPV at 9-10 years.
* Practice must have at least 100 eligible patients age 9-13 years

Exclusion Criteria:

* Practices with less than 100 eligible patients age 9-13 years
* Practices currently routinely recommend HPV vaccine at 9-10 years.
* Practices where less than 60% of providers agree to participate in the study.

Patient Eligibility Criteria

* Patient age 9-13 years
* Seen at a participating practice in the last 3 years
* Due for at least 1 dose of HPV vaccine

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3100 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Age at completion of two dose HPV series | post-intervention assessed in year 5 of study, year 4 of trial
  The primary outcome will be age at completion of the two dose HPV series. This is a time-to-event outcome, with the event of interest being vaccine completion. Comparisons between the intervention practices and control practices will be made. Practice electronic health records will be used to assess this outcome.

SECONDARY OUTCOMES:
HPV completion by age 13 years | post-intervention assessed in year 5 of study, year 4 of trial
  Secondary outcome will be HPV series completion rates by age 13. This will be a binary outcome. Comparisons between the intervention practices and control practices will be made. Practice electronic health records will be used to assess this outcome.
Age at initiation of the HPV series | post-intervention assessed in year 5 of study, year 4 of trial
  This is a time-to-event outcome, with the event of interest being vaccine initiation. Comparisons between the intervention practices and control practices will be made. Practice electronic health records will be used to assess this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of California at Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Yes
The study team guarantees that any and all data collected as part of this project will be released in accordance with standard data sharing policies and procedures to validate research findings if requested. Data will be made available in a timely manner to the broader scientific community, and will be complete, and as accurate as possible. All data released will be de-identified, with no information that could be linked to any study subjects, or participating study practices in order to ensure the confidentiality of all subjects and practices. If necessary, a data use agreement will be established.
Supporting Information: Study Protocol, SAP
Time Frame: May 2025
Access Criteria: The study team intends to share study data that may be requested from other research investigators in a data-sharing agreement provided at the individual study's end. The data-sharing agreement will include requirements to protect participants' privacy and data confidentiality. It will prohibit the recipient from transferring the data to other users and will require that the data's security be protected by standard means and be used for research purposes only. The method of distribution will be by request to Dr. Kempe (UCAMC) or Dr. Szilagyi (UCLA), the study PIs. After a requestor completes the data-sharing agreement, we will upload data to a secure File Transfer Protocol (FTP) site with the limited dataset to the requestor, or email the data through our University secured email systems that require users to create an account and sign-in with a username and password in order to receive and download any type of sensitive data.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04722822/SAP_000.pdf